CLINICAL TRIAL: NCT01041872
Title: Dose-effect of Propofol for Anesthetic Induction: Double-blind Comparison of Different Propofol Formulations Administered Alone or With Lidocaine
Brief Title: Comparison of Different Propofol Formulations
Acronym: Propofols
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009/22
Record Dates: First submitted 2009-12-31; First posted 2010-01-01 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: General Anesthesia
MeSH Terms: interventions — Lidocaine; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Propofol Astrazeneca (Active Comparator): Propofol with saline is administered using a closed-loop algorithm which permits to reach a Bispectral Index target of 50. The blinded syringe contains 45 ml of propofol and 5 ml of saline.
  Interventions: Drug: Propofol Astrazeneca plain
- Propofol Astrazeneca plus lidocaine (Experimental): Propofol with lidocaine 1¨% is administered using a closed-loop algorithm which permits to reach a Bispectral Index target of 50. The blinded syringe contains 45 ml of propofol and 5 ml of lidocaine.
  Interventions: Drug: Propofol Astrazeneca plus lidocaine
- Propofol-lipuro B. Braun plain (Experimental): Propofol with saline is administered using a closed-loop algorithm which permits to reach a Bispectral Index target of 50. The blinded syringe contains 45 ml of propofol and 5 ml of saline.
  Interventions: Drug: Propofol-lipuro B. Braun plain
- Propofol-lipuro B. Braun plus lidocaine (Experimental): Propofol with lidocaine 1¨% is administered using a closed-loop algorithm which permits to reach a Bispectral Index target of 50. The blinded syringe contains 45 ml of propofol and 5 ml of lidocaine.
  Interventions: Drug: Propofol-lipuro B. Braun plus lidocaine
- Propofol Fresenius plain (Experimental): Propofol with saline is administered using a closed-loop algorithm which permits to reach a Bispectral Index target of 50. The blinded syringe contains 45 ml of propofol and 5 ml of saline.
  Interventions: Drug: Propofol Fresenius plain
- Propofol Fresenius plus lidocaine (Experimental): Propofol with lidocaine 1¨% is administered using a closed-loop algorithm which permits to reach a Bispectral Index target of 50. The blinded syringe contains 45 ml of propofol and 5 ml of lidocaine.
  Interventions: Drug: Propofol Fresenius plus lidocaine

INTERVENTIONS:
Drug: Propofol Astrazeneca plain — Propofol with saline is administered using a closed-loop algorithm which permits to reach a Bispectral Index target of 50. The blinded syringe contains 45 ml of propofol and 5 ml of saline.
  Other Names: Propofol Astrazeneca
  Arms: Propofol Astrazeneca
Drug: Propofol Astrazeneca plus lidocaine — Propofol with lidocaine 1¨% is administered using a closed-loop algorithm which permits to reach a Bispectral Index target of 50. The blinded syringe contains 45 ml of propofol and 5 ml of lidocaine.
  Other Names: Propofol Astrazeneca, Lidocaine
  Arms: Propofol Astrazeneca plus lidocaine
Drug: Propofol-lipuro B. Braun plain — Propofol with saline is administered using a closed-loop algorithm which permits to reach a Bispectral Index target of 50. The blinded syringe contains 45 ml of propofol and 5 ml of saline.
  Other Names: Propofol-lipuro B. Braun
  Arms: Propofol-lipuro B. Braun plain
Drug: Propofol-lipuro B. Braun plus lidocaine — Propofol with lidocaine 1¨% is administered using a closed-loop algorithm which permits to reach a Bispectral Index target of 50. The blinded syringe contains 45 ml of propofol and 5 ml of lidocaine.
  Other Names: Propofol-lipuro B. Braun, lidocaine
  Arms: Propofol-lipuro B. Braun plus lidocaine
Drug: Propofol Fresenius plain — Propofol with saline is administered using a closed-loop algorithm which permits to reach a Bispectral Index target of 50. The blinded syringe contains 45 ml of propofol and 5 ml of saline.
  Other Names: Propofol Fresenius
  Arms: Propofol Fresenius plain
Drug: Propofol Fresenius plus lidocaine — Propofol with lidocaine 1¨% is administered using a closed-loop algorithm which permits to reach a Bispectral Index target of 50. The blinded syringe contains 45 ml of propofol and 5 ml of lidocaine.
  Other Names: Propofol Fresenius, lidocaine
  Arms: Propofol Fresenius plus lidocaine

SUMMARY:
The objective of this study is to evaluate the influence of different propofol formulations(plain or with lidocaine)on anesthetic induction. Propofol plain or with lidocaine is administered using a closed-loop algorithm in order to reach a Bispectral Index target of 50.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for an intravenous induction of anesthesia with propofol

Exclusion Criteria:

* Age under 18
* Pregnancy or breastfeeding
* Allergy to propofol, soya or peanuts,
* Allergy to lidocaine,
* History of central neurological disorder or brain injury,
* Patients receiving psychotropic drugs,
* Patient with a pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2009-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
necessary dose of propofol to obtain the induction of anesthesia (defined by a bispectral index of 50) | end of anesthetic induction

SECONDARY OUTCOMES:
calculated concentrations of propofol at the end of the anesthetic induction | end of the anesthetic induction
measured plasma propofol concentrations at the end of anesthetic induction (in 20% of patients) | 3 months after the end of patient's recruitment
pain at injection | during the PACU (post-anaesthesia care unit) stay
heart rate and arterial pressure modifications induced by anesthetic induction | end of anesthetic induction
patients satisfaction | during the PACU stay
necessary dose of propofol to obtain loss of consciousness | end of anesthetic induction
calculated concentrations of propofol at loss of consciousness | end of anesthetic induction

CONTACTS AND LOCATIONS:
Overall Officials: Morgan LeGuen, MD, Principal Investigator — Hôpital Foch
Locations (3):
- France (3):
  - Clinique Saint Augustin, Bordeaux
  - Laboratoire de Pharmacologie Toxicologie, hôpital Raymond Poincaré, Garches
  - Hôpital Foch, Suresnes

REFERENCES:
- [Background] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963